CLINICAL TRIAL: NCT00282282
Title: Tacrolimus and Sirolimus as Graft Versus Host Disease Prophylaxis After Allogeneic Non-myeloablative Peripheral Blood Stem Cell Transplantation
Brief Title: Tacrolimus and Sirolimus as Prophylaxis After Allogenic Non-myeloablative Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-362
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-03

CONDITIONS: Graft Versus Host Disease; GVHD
Keywords: non-myeloablative peripheral blood stem cell; PBSCT; tacrolimus; sirolimus
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Sirolimus; fludarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tacrolimus — Given orally just prior to and following stem cell transplant
Drug: sirolimus — Given orally just prior to and following stem cell transplant
Drug: fludarabine — Given once daily over 30 minutes for 4 days
Drug: busulfex — Given intravenously over 3 hours for 4 days

SUMMARY:
The purpose of this study is to extend the use of Tacrolimus and Sirolimus to determine how effective it is in preventing graft versus host disease (GVHD)in patients that have received non-myeloablative peripheral blood stem cell transplantation.

DETAILED DESCRIPTION:
* After the screening procedures confirm that the patient is eligible to participate in the research study, they will be admitted to the hospital to receive chemotherapy and stem cell transplantation (SCT). The duration of the hospitalization for the procedure is approximately 8 days.
* Patients will receive fludarabine once daily over 30 minutes intravenously for 4 days and busulfex once daily over 3 hours intravenously each day for the same 4 days.
* Just prior to the transplant and following the transplant the patient will receive sirolimus and tacrolimus to help prevent Graft versus Host Disease (GvHD). Both medications are taken orally.
* Patients will also take medications to help prevent possible infections (e.g. acyclovir). Filgrastim, a white blood cell growth factor, will be given daily in an injection under the skin, starting the day after the stem cell transplant and until the patients blood counts have recovered.
* After the stem cell infusion, the patient will be examined and have blood tests weekly for 1 month. At about the 1-month visit, a bone marrow biopsy and/or blood tests will be performed to determine the percentage of donor's cells in the blood or bone marrow. These tests will be repeated at 3-4 months after transplant.
* At 3-4 months after the transplant, patients will also have tests to reassess the response of your disease to transplant. This may involve a bone marrow biopsy, blood tests, and/or radiology studies depending upon the type of cancer.
* Follow-up will continue for the remainder of the patients life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies who are at a high risk of complications after conventional transplantation
* Availability of a related donor who is identical at 6 HLA loci
* Greater than 18 years of age
* Performance status 0-2
* Life expectancy of > 100 days

Exclusion Criteria:

* Pregnancy
* Evidence of HIV infection
* Heart failure uncontrolled medication
* Total bilirubin > 2.0mg/dl that is due to hepatocellular dysfunction
* AST >90
* Serum Creatinine >2.0
* Cholesterol > 300mg/dl while adequately treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Ho VT, Aldridge J, Kim HT, Cutler C, Koreth J, Armand P, Antin JH, Soiffer RJ, Alyea EP. Comparison of Tacrolimus and Sirolimus (Tac/Sir) versus Tacrolimus, Sirolimus, and mini-methotrexate (Tac/Sir/MTX) as acute graft-versus-host disease prophylaxis after reduced-intensity conditioning allogeneic peripheral blood stem cell transplantation. Biol Blood Marrow Transplant. 2009 Jul;15(7):844-50. doi: 10.1016/j.bbmt.2009.03.017. PMID 19539216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with hematologic malignancies who were at high risk of complications after conventional transplantation, with 6/6 HLA matched-related donors were approached with information about participating in the study. Participants were approached at either inpatient or outpatient clinics by physicians between 2006 and 2007.
Groups:
- Tacrolimus and Sirolimus: Participants received a tacrolimus and sirolimus graft-versus-host disease (GVHD) prophylaxis regimen. Tacrolimus was given 0.05 mg/kg/day (in 2 daily divided doses) orally starting 3 days before bone marrow transplant with a target serum concentration of 5-10ng/mL. Sirolimus was administered with a 12mg oral loading dose 3 days prior to transplantwith a target serum concentration of 3-12ng/mL. Tapering of tacrolimus and sirolimus doses was encouraged starting 64 days after transplant with a goal of discontinuing immunosuppression therapy approximately 6 months after transplant if there were no signs of GVHD.
Period: Overall Study
Arm/Group | Tacrolimus and Sirolimus
Started | 29 (31 patients enrolled but 2 patients did not go through with transplant)
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus and Sirolimus
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 53 [29 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade II-IV Acute GVHD (aGVHD) Developing by Day 100 Following Non-myeloablative PBSC Transplantation Using Tacrolimus and Sirolimus.
Description: All participants received tacrolimus and sirolimus in this one arm study. There were no participants considered unevaluable for this measure (deceased prior to day 100). The total number of people who developed grade II-IV aGVHD before day 100 are reported here.
Time Frame: 100 days
Population: Participants who lived more than 30 days posttransplant were considered evaluable. Incidence of grade II-IV aGVHD was adjusted for participants who had aGVHD off-treatment.
Measure: Number; unit: participants
Arm/Group | Tacrolimus and Sirolimus
Number analyzed (Participants) | 29
participants | 5

2. Secondary Outcome: Percentage of Participants With ≥90 Percent Donor-derived Hematopoeisis Around 100 Days Post Transplantation
Description: The percentage of participants with ≥90 percent donor-derived hematopoeisis was assessed around day +100 using peripheral blood chimerism.
Time Frame: 100 days
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus and Sirolimus
Number analyzed (Participants) | 27
percentage of participants | 78 [11 to 100]

3. Secondary Outcome: Disease Response.
Description: Disease response was assessed as 2 year progression-free survival. The median follow-up time was 1.84 years. The percentage of participants with who reached this timepoint with no disease progression are reported.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus and Sirolimus GVHD Prophylaxis
Number analyzed (Participants) | 29
percentage of participants | 48 [29 to 64]

ADVERSE EVENTS:
Time Frame: Participants were followed for approximately 2 years post-transplant
Arm/Group | Tacrolimus and Sirolimus
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus and Sirolimus (N=29)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1 — 1 patient had transplantation-associated thrombotic microangiopathy that resolved with the discontinuation of tacrolimus

LIMITATIONS AND CAVEATS:
This study is a single-institution study, and as such the data are limited by the small study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No